CLINICAL TRIAL: NCT06515535
Title: Efficacy of Topical Tranexamic Acid in Reducing Blood Loss During Elective Cesarean Delivery in Patients With Placenta Previa
Brief Title: Efficacy of Topical Tranexamic Acid in Reducing Blood Loss During CS in Patients With Placenta Previa
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdalla Mousa, Lecturer of obgyn Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MS-201-2024
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Placenta Previa
MeSH Terms: conditions — Placenta Previa | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (n=28) (Experimental): The topical tranexamic acid group will receive topical tranexamic acid after placental delivery applied on the placental bed for 5 minutes by using a sterile towel soaked with 2g tranexamic acid (Kapron, Amoun, Cairo, Egypt) (4 ampules 500ug) diluted in 100ml of sodium chloride 0.9%, in addition to the IV infusion of 1g tranexamic acid (2 ampules 500ug) diluted with 20ml of 5% glucose administered just after delivery of the fetus.
  Interventions: Drug: Topical tranexamic acid; Drug: Intravenous tranexamic acid
- Control group (n=28) (Active Comparator): The intravenous tranexamic acid group will receive only an IV infusion of 1g of tranexamic acid (2 ampules 500ug) diluted with 20 ml of 5% glucose administered just after delivery of the fetus.
  Interventions: Drug: Intravenous tranexamic acid

INTERVENTIONS:
Drug: Topical tranexamic acid — Topical tranexamic acid will be applied after placental delivery on the placental bed for 5 minutes by using a sterile towel soaked with 2g tranexamic acid (Kapron, Amoun, Cairo, Egypt) (4 ampules 500ug) diluted in 100ml of sodium chloride 0.9%
  Arms: Study group (n=28)
Drug: Intravenous tranexamic acid — Intravenous tranexamic acid will be given in the form of an IV infusion of 1g of tranexamic acid (2 ampules 500ug) diluted with 20 ml of 5% glucose administered just after delivery of the fetus.

SUMMARY:
Objectives: To evaluate the efficacy of topical tranexamic acid applied on the placental bed after placental delivery to reduce blood loss during cesarean delivery in women with placenta previa.

Patients will be randomly assigned into two groups:

Group (A) - Study group (n=28): The topical tranexamic acid group will receive topical tranexamic acid after placental delivery applied on the placental bed for 5 minutes by using a sterile towel soaked with 2g tranexamic acid (Kapron, Amoun, Cairo, Egypt) (4 ampules 500ug) diluted in 100ml of sodium chloride 0.9%, in addition to the IV infusion of 1g tranexamic acid (2 ampules 500ug) diluted with 20ml of 5% glucose administered just after delivery of the fetus.

Group (B) - Control group (n=28): The intravenous tranexamic acid group will receive only an IV infusion of 1g of tranexamic acid (2 ampules 500ug) diluted with 20 ml of 5% glucose administered just after delivery of the fetus.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-40 years old.
* BMI less than 30 kg/m2.
* Pregnancy of singleton living fetus.
* Placenta previa by ultrasound assessment
* Gestational age > 36 weeks.

Exclusion Criteria:

* Women with a history of any medical disorder with pregnancy, e.g., Gestational diabetes and hypertension.
* Women with systemic diseases, e.g., diabetes mellites, systemic immune disorders such as systemic lupus erythematosus
* Women with bleeding tendency or coagulopathy.
* Women on anticoagulants or hemodynamically unstable women.
* Women with uterine abnormalities, such as fibroids or polyps.
* Emergency termination of pregnancy.
* Intrauterine fetal death.
* Pregnancy with obstetric hemorrhage, e.g., antepartum hemorrhage
* Cases of placenta accrete spectrum disorder or placental abruption
* Women with known allergies to Tranexamic acid

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-07-24 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Amount of blood loss | during operation
  amount of intraoperative blood loss during CS in patients with placenta previa

SECONDARY OUTCOMES:
operative time | during operation